CLINICAL TRIAL: NCT02988765
Title: Ultrasound Morphometric and Cyto/Histological Combined Pre-operative Assessment of Inguinal Lymph Node Status in Women With Invasive Vulvar Carcinoma
Acronym: Morpho-Node
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Morpho-Node
Record Dates: First submitted 2016-12-02; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Vulvar Cancer
Keywords: vulvar cancer; inguinal lymph node; lymph node status; cytology; core biopsy
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Invasive vulvar cancer (IVC) (Experimental): * Vulvar carcinoma (stromal infiltration > 1 mm)
  * Histotypes different from squamous cells carcinomas are included
  Interventions: Procedure: Groin ultrasound +/- fine needle aspiration

INTERVENTIONS:
Procedure: Groin ultrasound +/- fine needle aspiration — Preoperative ultrasound morphometry (USM) of the inguino-femoral lymph nodes (IFLN).
  The FNAC and/or FNAB is performed in case of suspicious nodes, if at least one of the selected criteria is relieved during ultrasound

SUMMARY:
Vulvar cancer is a rare and very aggressive cancer, mainly spreading through lymphatics, in which the preoperative evaluation is critical to address surgery between sentinel node biopsy or radical groin lymphadenectomy.

DETAILED DESCRIPTION:
In the absence of clearly an specific guidelines on preoperative vulvar cancer assessment, the investigators decided to better investigate the role of ultrasound in groin nodes evaluation through the study 10 sonographic features of suspicion for nodal involvement:

* globular shape (loss of the normal elliptical form)
* long/short axis ratio
* cortical/medulla ratio
* cortical focal bulging or thickening
* hilum anomalies
* inhomogeneous echostructure
* intranodal deposits
* extracapsular spread
* grouping
* vascularization

The standard of comparison is histopathology.

The prospectively evaluation of these parameters will be obtained on the enrolled patients.

The investigators also provided the retrospective review - by specialized staff - of ultrasound images collected in archives associated with information relating to the cyto/histological procedures (performed in case of suspicious lymph nodes) in patients who underwent surgical treatment in the last five years at the study center.

ELIGIBILITY:
Inclusion Criteria:

* Invasive vulvar cancer (all infiltrating histotypes)
* Age >18 years

Exclusion Criteria:

* patient unable to follow the study procedures
* patient with major depressive disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy, negative predictive value (NPV) and positive predictive value (PPV) of ultrasound morphometry (USM) in the prediction of groin lymph node status | within the first 30 days after surgery
Accuracy, negative predictive value (NPV) and positive predictive value (PPV) of fine needle aspiration in the prediction of groin lymph node status | within the first 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gynecologic Oncology/Fondazione Policlinico Gemelli, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No